CLINICAL TRIAL: NCT03220399
Title: Pharmacokinetic Interaction and Safety/Tolerability Between NVP-1603-1 and NVP-1603-2 in Healthy Male Volunteers
Brief Title: Pharmacokinetic Interaction and Safety/Tolerability Between NVP-1603-1 and NVP-1603-2
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Decided to stop drug development
Sponsor: NVP Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NVP-1603_P1_DDI
Record Dates: First submitted 2017-06-30; First posted 2017-07-18 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NVP-1603-1 (P) (Experimental): Drug: NVP-1603-1
  1capsule, oral dosing
  Interventions: Drug: NVP-1603-1 (P)
- NVP-1603-2(T) (Experimental): Drug: NVP-1603-2
  1Tablet, oral dosing
  Interventions: Drug: NVP-1603-2 (T)
- NVP-1603-1and NVP-1603-2 (P+T) (Experimental): Drug: NVP-1603-1, 1capsule and NVP-1603-2, 1Tablet co-adminstration (oral dosing)
  Interventions: Drug: NVP-1603-1 and NVP-1603-2 (P+T)

INTERVENTIONS:
Drug: NVP-1603-1 (P) — 1capsule, single oral dosing
  Other Names: NVP-1603-1
  Arms: NVP-1603-1 (P)
Drug: NVP-1603-2 (T) — 1tablet, single oral dosing
  Other Names: NVP-1603-2
  Arms: NVP-1603-2(T)
Drug: NVP-1603-1 and NVP-1603-2 (P+T) — 1capsule and 1tablet co-administration, oral single dosing
  Other Names: NVP-1603-1 and NVP-1603-2
  Arms: NVP-1603-1and NVP-1603-2 (P+T)

SUMMARY:
The purpose of this study is to compare the pharmacokinetics and safety/tolerability between NVP-1603-1 and NVP-1603-2

DETAILED DESCRIPTION:
pharmacokinetics and safety/tolerability between NVP-1603-1 and NVP-1603-2

ELIGIBILITY:
Inclusion Criteria:

* Men 19years of age or older at screening test.
* BMI of >18.5kg/㎡ and <27.0kg/㎡ subject, weight more than 50kg.
* Subject has signed and dated informed consent.

Exclusion Criteria:

* Treatment with an investigational product (Phase I study or Biological study) within 3month preceeding the first dose of study medication.
* History of (or presence) study medication absortion, distribution, metabolism(e.g., liver/ductal, kidney, cardio-vascular, endocrine, respiratory, GI, hematology, oncology, CNS, musculo-skeletal) or related past medical/surgery history
* Current alcohol abuse.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy males (19years of age or older)
Enrollment: 0 (Actual)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-03-28 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic interaction | 0h - 48hrs
  Area under the curve (AUC)

IPD SHARING:
Plan to Share IPD: Undecided